CLINICAL TRIAL: NCT00766545
Title: Cilostazol Stroke Prevention Study : A Placebo-controlled Double-blind Trial for Secondary Prevention of Cerebral Infarction.
Acronym: CSPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 021-91-001
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cilostazol (Experimental): cilostazol oral tablet 100 mg, twice daily
  Interventions: Drug: cilostazol
- placebo (Placebo Comparator): placebo of cilostazol, twice daily
  Interventions: Drug: placebo of cilostazol

INTERVENTIONS:
Drug: cilostazol — oral tablet 100 mg, twice daily, over 1 year
  Arms: cilostazol
Drug: placebo of cilostazol — oral tablet, 0 mg twice daily, over 1 year
  Arms: placebo

SUMMARY:
The multi-center, double-blind, placebo-controlled, randomized, group-comparison study was designated to assess the long-term safety and efficacy of the antiplatelet drug cilostazol in preventing the recurrence of cerebral infarction in patients who had suffered a cerebral infarction 1 to 6 months prior to entering the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Prior cerebral infarction Onset at 1 to 6 months before randomization
2. CT or MRI detection of responsible site
3. Without serious complications (malignant tumor, liver cirrhosis, renal failure, or heart failure)

Exclusion Criteria:

1. History of intracranial hemorrhage
2. Possibility of cardiogenic cerebral embolism in the past or future All patients with any of the following complications were excluded: mitral valve stenosis, prosthetic valve, endocarditis, myocardial infarction within 6 weeks after onset, ventricular aneurysm, intraventricular or intraatrial blood clots, mitral valve prolapsed (age under 45 years old, lacking other causes for cerebral embolism induction), atrial fibrillation, sick sinus syndrome, idiopathic cardiomyopathy
3. Severe cerebral deficits rendering the patient bed-ridden, totally dependent, or demented
4. Contraindications to the study drug Hemostatic disorders or systemic bleeding Pregnant or possibly pregnant women, or nursing mothers
5. Requirement for nonstudy antiplatelet drugs, anticoagulant drugs, or fibrinolytic drugs for another disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 1992-04; Primary Completion 1997-03 (Actual); Study Completion 1997-03 (Actual)

PRIMARY OUTCOMES:
Recurrence of cerebral infarction | any time

SECONDARY OUTCOMES:
Cerebral infarction or myocardial infarction, Cerebral infarction, intracranial hemorrhage, or TIA, Cerebral infarction, intracranial hemorrhage, myocardial infarction, or vascular death, All vascular events, vascular death, and Death from any cause | any time

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto Area, Japan